CLINICAL TRIAL: NCT06743659
Title: Alert-Based Computerized Decision Support for Identification and Management of Patients With Familial Hypercholesterolemia (FH-ALERT Trial)
Brief Title: Computerized Decision Support for Identification and Management of Familial Hypercholesterolemia
Acronym: FH-ALERT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gregory Piazza, MD, MS, Staff Physician, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024P001619
Record Dates: First submitted 2024-12-18; First posted 2024-12-20 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Familial Hypercholesterolaemia
Keywords: Familial Hypercholesterolemia; Computerized Decision Support; Electronic Alerts; High Cholesterol
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: During the first 6 months, the BPA will run in "silent mode" and will not provide notification to the clinician of record about the potential diagnosis of FH. For the following 18 months, the BPA will run in "alert mode" during which an on-screen alert will notify the ambulatory care clinician of record that the patient has a "definite," "probable," or "possible" diagnosis of FH but has not been recognized as such.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pre-Alert (No Intervention): In the Pre-Alert phase of 6 months, patients meeting enrollment criteria will be identified but the clinician will not be notified regarding the possible diagnosis of Familial Hypercholesterolemia.
- Alert (Experimental): In the Alert phase of 18 months, an on-screen alert through the Electronic Health Record will notify the ambulatory care clinician of record that the patient has a "definite," "probable," or "possible" diagnosis of FH but has not been recognized as such.
  Interventions: Device: Alert-based computerized decision support

INTERVENTIONS:
Device: Alert-based computerized decision support — A program will be designed to run within the Electronic Health Record (EHR) that will identify outpatients with "definite," "probable," or "possible" diagnosis of FH. The BPA will calculate the Dutch Lipid Clinic Network score using the following EHR data:
  1. Maximum LDL-C level in the laboratory results
  2. Abnormal genetic testing for FH in the laboratory results
  3. Medical history or problem list entry for tendinous xanthomata or arcus cornealis
  4. Medical history, visit diagnosis, or problem list entry of premature CAD, cerebrovascular disease, or PAD
  5. Family history of premature CAD, cerebrovascular disease, or PAD
  In the Alert phase, an on-screen alert will notify the ambulatory care clinician of record that the patient has a "definite," "probable," or "possible" diagnosis of FH. ambulatory care clinician will have the opportunity to proceed to an order template through which a referral for specialty care focused on evaluation and management of FH can be made.
  Other Names: Best Practice Advisory; Computer Alert
  Arms: Alert

SUMMARY:
The goal of this clinical trial is to learn if a computer alert can aid clinicians in identifying patients with a genetic type of high cholesterol, called Familial Hypercholesterolemia. The main question it aims to answer is whether the computer alert increases recognition of this high cholesterol disorder.

DETAILED DESCRIPTION:
FH-ALERT is a single-center, time-series trial of a patient- and provider-facing EPIC BPA (alert-based CDS tool) to increase diagnosis, LDL-C lowering, and guideline-based therapy of outpatients with presentations consistent with FH. For the first 6 months, the BPA will run in "silent mode", identifying patients with presentations consistent with FH, but not alerting the clinician of record. Following this initial "pre-alert" 6-month period, the BPA will switch to "alert mode" for 18 months, which will provide the on-screen notification to the clinician of record. In other words, consecutive outpatients with presentations consistent with FH will be enrolled over two years: "pre-alert" (silent mode) for 6 months and "alert mode" for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* seen in the BWH Endocrinology, Cardiovascular Medicine, and Primary Care Clinics
* Dutch Lipid Clinic Network score of at least 3 points

Exclusion Criteria:

* a Familial Hypercholesterolemia diagnosis already documented in the EHR medical history, visit history, or problem list

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of documented FH diagnosis | 6 Months
  We will review the medical history, visit diagnosis, and problem list sections of the Electronic Health Record (EPIC) to make this determination of diagnosis of Familial Hypercholesterolemia.

SECONDARY OUTCOMES:
Mean Change in LDL-C | 6 Months
  Mean change in LDL-C levels within 6 months following triggering of the BPA compared with the most recent LDL-C prior to the clinic visit in outpatients with presentations consistent with FH ("definite," "probable," or "possible" Dutch Lipid Clinic Network score).

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Will provide data upon reasonable request after publication of study.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: After completion of the study for a period of 10 years
Access Criteria: Investigators with a scientifically sound reason for accessing the data upon reasonable request